CLINICAL TRIAL: NCT04082221
Title: The Influence of Different Sample Collection and DNA Extraction Methods on the Bacterial Composition of the Gut of Healthy Subjects
Brief Title: Comparison of Different Methods for the Analysis of Gut Microbiome Composition
Acronym: COLLECT
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Dr. Lajos Marko, Principal Investigator, Charite University, Berlin, Germany
Other Study IDs: ChariteU-ECRC-COLLECT
Record Dates: First submitted 2019-09-05; First posted 2019-09-09 (Actual); Last update posted 2019-09-11 (Actual); Status verified 2019-09

CONDITIONS: Healthy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Stool (stool DNA), Blood Serum and Blood Plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
The human gastrointestinal tract shelters a complex and dynamic population of microorganisms, the gut microbiota, which plays an important role in immune and metabolic homeostasis. In recent years several major diseases were linked with alterations in the gut microbiome composition.

There are known factors which can influence gut microbiata composition. For example diet is known to play a fundamental role in determining the composition of the intestinal microbiota over time. However, there are very few studies evaluating how collection and DNA isolation methods affect microbiome composition.

DETAILED DESCRIPTION:
An observational clinical study with 28 healthy subjects is planned to assess how different commercially available stool sampling kits and fecal DNA extraction kits influence the apparent composition of the gut microbiome. Participants will be instructed to collect stool samples at two time points separated by one week using six different methods (naïve and Zymo DNA/RNA Shield kit on dry ice as well as OMNIgene GUT, RNALater, 95% EtOH, Zymo DNA/RNA Shield at room temperature). DNA extraction from all samples will be performed using QIAamp Power Fecal (Qiagen, N. V) and ZymoBIOMICS (Zymo Research, CA.).

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-60
* Body mass index (BMI) 18,5- 29,9 kg/m2
* Willingness to participate in the study examination and fecal sample collection process

Exclusion Criteria:

* Subjects currently on medication (with the exception of contraceptives)
* Subjects with acute or chronic disease
* Pregnant or lactating women
* Subjects with a history of drug or alcohol abuse
* Subjects on a vegan diet
* Subjects who are legal incapacitated or their circumstances do not enable the patient to fully understand the nature, significance and scope of this study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy subjects
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2019-03-11 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-09-05 (Actual)

PRIMARY OUTCOMES:
Collection of stool samples | one week
  Collection of 2 stool samples in one week using different conditions
  DNA extraction from all samples will be performed using QIAamp Power Fecal (Qiagen, N. V) and ZymoBIOMICS (Zymo Research, CA.) to assess how different commercially available stool sampling kits and fecal DNA extraction kits influence the apparent composition of the gut microbiome

CONTACTS AND LOCATIONS:
Overall Officials: Anja Mähler, PhD, Study Chair — Franz-Volhard-Centr. at the Experimental and Clinicial Research Center
Locations (1):
- Experimental and Clinical Research Center, Clinical Research Unit, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hart ML, Meyer A, Johnson PJ, Ericsson AC. Comparative Evaluation of DNA Extraction Methods from Feces of Multiple Host Species for Downstream Next-Generation Sequencing. PLoS One. 2015 Nov 24;10(11):e0143334. doi: 10.1371/journal.pone.0143334. eCollection 2015. PMID 26599606
- [Background] Wesolowska-Andersen A, Bahl MI, Carvalho V, Kristiansen K, Sicheritz-Ponten T, Gupta R, Licht TR. Choice of bacterial DNA extraction method from fecal material influences community structure as evaluated by metagenomic analysis. Microbiome. 2014 Jun 5;2:19. doi: 10.1186/2049-2618-2-19. eCollection 2014. PMID 24949196